CLINICAL TRIAL: NCT00830518
Title: A Phase 2 Trial of MLN8237, an Oral Aurora A Kinase Inhibitor, in Adult Patients With Acute Myelogenous Leukemia and High-Grade Myelodysplastic Syndrome
Brief Title: A Phase 2 Trial of MLN8237 in Adult Participants With Acute Myelogenous Leukemia and High-Grade Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C14005; 2008-006977-34 (EudraCT Number); U1111-1187-6569 (Registry Identifier: WHO)
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Acute Myelogenous Leukemia; High-Grade Myelodysplastic Syndrome
Keywords: Drug therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alisertib (Experimental): Alisertib 50 mg, capsules, orally, twice daily for 7 days, followed by 14-day washout period, in 21-day cycles until disease progression or unacceptable treatment-related toxicity (Up to 26 Cycles).
  Interventions: Drug: Alisertib

INTERVENTIONS:
Drug: Alisertib — Alisertib capsules
  Other Names: MLN8237

SUMMARY:
This is an open-label, multicenter, phase 2 study of alisertib (MLN8237) in participants with acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
The drug being tested in this study is called alisertib (MLN8237). Alisertib is being tested to treat people who have acute myeloid leukemia (AML) or high-grade myelodysplastic syndrome (MDS). This study looked at the antitumor activity in people who received alisertib.

The study enrolled 57 patients. Participants were categorized by disease sub-types AML and MDS. Participants received:

• Alisertib 50 mg

All participants took alisertib capsules every 12 hours each day for 7 days followed by a 14-day rest period in 21-day cycles for approximately 26 cycles.

This multi-center trial was conducted in North America and France. The overall time to participate in this study was until there is evidence of disease progression or unacceptable treatment-related toxicity. The participant could continue treatment beyond 12 months if it was considered by the Sponsor and the Investigator that they would derive benefit from continued alisertib treatment. Participants had weekly blood work and clinic visits, with disease assessments every 2 cycles (ie. every 6 weeks) up to and including Cycle 16. Reduced visits (every 12 weeks) were conducted for participants tolerating treatment beyond Cycle 16 and for participants off treatment without disease progression.

ELIGIBILITY:
Inclusion Criteria:

Each participants must meet all of the following inclusion criteria:

1. Male or female participants 18 years or older
2. Eligible diagnoses:

   * Acute myelogenous leukemia (except acute promyelocytic leukemia [APL]) with > 10% bone marrow or peripheral blood blasts; failed to achieve complete response (CR) or relapse after prior therapy, not candidates for potentially curative treatment. Untreated participants > 60 are eligible if not candidates for standard induction.
   * High-grade myelodysplastic syndrome (MDS), defined by all the following features: International Prognostic Scoring System (IPSS) Intermediate-2 or High Risk; > 10% blasts on bone marrow examination; treatment failure from, or not candidates for, standard therapies including demethylating agents, e.g. azacytidine or decitabine.
3. Eastern Cooperative Oncology Group performance status 0-2
4. Female participants:

   * Postmenopausal for at least one year
   * Surgically sterile, or
   * If childbearing potential, agree to practice two effective methods of contraception or abstain from heterosexual intercourse.
5. Male participants:

   * Practice effective barrier contraception to one month after the last dose of study drug, or
   * Abstain from heterosexual intercourse.
6. Voluntary written consent
7. Participants on hydroxyurea may be included

Exclusion Criteria:

1. Pregnant or lactating females
2. Known human immunodeficiency virus (HIV) positive or acquired immune deficiency syndrome (AIDS) - related illness
3. Serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the protocol completion
4. Total bilirubin > 1.5 × the upper limit of normal (ULN)
5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5 × the ULN. AST, ALT may be elevated to 5 x the ULN if reasonably ascribed to underlying hematological disorder.
6. Calculated creatinine clearance < 30 mL/minute
7. Antineoplastic or radiotherapy within 14 days preceding the first dose
8. Myocardial infarction within 6 months of enrollment or current history of New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia
9. Major surgery 14 days prior to the first dose
10. Clinically uncontrolled central nervous system (CNS) involvement.
11. Inability to swallow capsules
12. History of uncontrolled sleep apnea or conditions that result in excessive daytime sleepiness, such as chronic lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-02-10 (Actual); Primary Completion 2010-02-02 (Actual); Study Completion 2011-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Hematology and Oncology Associates of Northern New Jersey, Morristown, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 19 investigative sites in France, Canada and the United States from 10 February 2009 to 04 July 2011.
Pre-assignment Details: Participants with a diagnosis of acute myelogenous leukemia or myelodysplastic syndrome received 50 mg alisertib twice daily for 7 days in 21 day cycles. Results are reported according to lymphoma disease subtypes: acute myelogenous leukemia and myelodysplastic syndrome.
Groups:
- Alisertib 50 mg (Acute Myeloid Leukemia): Participants with acute myeloid leukemia received alisertib 50 mg, capsules, orally, twice daily for 7 days, followed by 14-day washout period, in 21-day cycles until disease progression or unacceptable treatment-related toxicity (Up to 26 Cycles).
- Alisertib 50 mg (Myelodysplastic Syndrome): Participants with myelodysplastic syndrome received alisertib 50 mg, capsules, orally, twice daily for 7 days, followed by 14-day washout period, in 21-day cycles until disease progression or unacceptable treatment-related toxicity (Up to 6 Cycles).
Period: Overall Study
Arm/Group | Alisertib 50 mg (Acute Myeloid Leukemia) | Alisertib 50 mg (Myelodysplastic Syndrome)
Started | 46 | 11
Completed | 0 (Completed = participants who completed study treatment.) | 0
Not Completed | 46 | 11
Not completed — Progressive Disease | 18 | 8
Not completed — Symptomatic Deterioration | 4 | 1
Not completed — Adverse Event | 14 | 1
Not completed — Withdrawal by Patient | 2 | 0
Not completed — Reason not Specified | 8 | 1

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all participants who received any amount of alisertib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alisertib 50 mg (Acute Myeloid Leukemia) | Alisertib 50 mg (Myelodysplastic Syndrome) | Total
Number analyzed (Participants) | 46 | 11 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (7.41) | 69.5 (12.50) | 71.4 (8.54)
Age, Customized [Number; unit: participants]
  <60 years | 4 | 2 | 6
  ≥60 years | 42 | 9 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 3 | 25
  Male | 24 | 8 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 34 | 9 | 43
  Not Reported | 10 | 2 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  White | 36 | 10 | 46
  Black or African American | 3 | 0 | 3
  Asian | 1 | 0 | 1
  Not Reported | 6 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 33 | 9 | 42
  France | 11 | 2 | 13
  Canada | 2 | 0 | 2
Height [Mean (Standard Deviation); unit: cm] — Population: Baseline height data is available for n=36,10 participants, respectively.
  cm
    number analyzed (Participants) | 36 | 10 | 46
    (all) | 165.8 (8.35) | 171.4 (9.98) | 167.0 (8.93)
Weight [Mean (Standard Deviation); unit: kg] — Population: Baseline weight data is available for n=45,11 participants, respectively.
  kg
    number analyzed (Participants) | 45 | 11 | 56
    (all) | 73.7 (13.80) | 80.4 (17.27) | 75.0 (14.62)
Baseline Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] — Population: Baseline BSA data is available for n=36,10 participants, respectively.
  m^2
    number analyzed (Participants) | 36 | 10 | 46
    (all) | 1.83 (0.203) | 1.94 (0.262) | 1.86 (0.219)
Years Since Initial Diagnosis [Mean (Standard Deviation); unit: years] | 0.65 (0.793) | 0.82 (0.780) | 0.68 (0.787)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG performance is defined as: 0=Normal activity (fully active, able to carry on all predisease performance without restriction); 1=Symptoms but ambulatory (restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature); 2=In bed <50% of the time (ambulatory and capable of all self-care, but unable to carry out any work activities.
  participants
    0 | 9 | 3 | 12
    1 | 29 | 8 | 37
    2 | 8 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (ORR) Based on Investigator's Assessment
Description: Best ORR is defined as the number of participants with complete remission(CR) or partial remission(PR) assessed by the Investigator using modified AML/MDS International Working Group(IWG) Criteria. AML:CR=neutrophils >1x10^9/L, platelets >100x10^9/L, bone marrow blasts(BMB) <5%, transfusion independent, no extramedullary disease(EMD); CRi=BMB <5%, transfusion independent, no EMD; PR=neutrophils >1x10^9/L, platelets >100x10^9/L, BMB >50% decrease and 5% to 25%, blasts <5% with Auer rods; PRi=BMB >50% decrease and 5% to 25%. MDS:CR=bone marrow: ≤5% myeloblasts with normal maturation, peripheral blood: hemoglobin ≥11 g/dL, platelets ≥100x10^9/L, neutrophils ≥1.0x10^9/L, blasts 0%; PR=all CR criteria if abnormal before treatment except: BMB decreased by ≥50% over pretreatment but still >5%; PRi=BMB decreased by ≥50% over pretreatment but still >5%; Marrow CR=bone marrow: ≤5% myeloblasts and decrease by ≥50% over pretreatment, peripheral blood hematologic improvement responses noted.
Time Frame: Baseline and every 2 cycles up to Cycle 16 (up to Month 12), from Cycle 17 every 4 cycles until disease progression, after end of treatment every 12 weeks for up to 12 Months (Approximately 2.4 years)
Population: Response-Evaluable Population included all participants who received at least 1 dose of alisertib and had at least 1 post-baseline response assessment. In 2 participants disease transformed from MDS to AML. One participant is considered AML and one participant is considered MDS in the calculation, based on the timing of their transformation.
Measure: Number; unit: participants
Arm/Group | Alisertib 50 mg (Acute Myeloid Leukemia) | Alisertib 50 mg (Myelodysplastic Syndrome)
Number analyzed (Participants) | 35 | 10
participants
  CR + PR | 6 | 0
  Complete Remission (CR + CRi + Marrow CRi) | 1 | 0
  Partial Remission (PR + PRi) | 5 | 0
  Stable Disease as Best Response | 17 | 2

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of first study drug administration to the date of first documented progressive disease (PD) or death.
Time Frame: as for outcome 1
Population: Response-Evaluable Population included all participants who received at least 1 dose of alisertib and had at least 1 post-baseline response assessment. For a participant that has not progressed and has not died, PFS is censored at the last response assessment that is SD or better.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alisertib 50 mg (Acute Myeloid Leukemia) | Alisertib 50 mg (Myelodysplastic Syndrome)
Number analyzed (Participants) | 35 | 10
days | 55.0 [47.0 to 67.0] | 38.0 [35.0 to 113.0]

3. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response is defined as the time from the date of first documentation of a response to the date of first documented PD.
Time Frame: as for outcome 1
Population: Response--Evaluable Population included all participants who had measurable disease, received at least 1 dose of alisertib, and had at least 1 post baseline response assessment. All responders were evaluated in this outcome measure. For a participant that has not progressed, DOR is censored at the last response assessment that is SD or better.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alisertib 50 mg (Acute Myeloid Leukemia) | Alisertib 50 mg (Myelodysplastic Syndrome)
Number analyzed (Participants) | 6 | 0
days | 409.0 [57.0 to 596.0] |

4. Secondary Outcome: Best Overall Hematologic Improvement (HI) Response for Myelodysplastic Syndrome Based on Investigator Assessment
Description: Best overall HI response is defined as percentage of participants with response as assessed by Investigator based on IWG criteria: 1)Erythroid response (pretreatment,<11 g/dL): hemoglobin (Hgb) increase by ≥1.5 g/dL, relevant reduction of units of red blood cell (RBC) transfusions by absolute number of at least 4 RBC transfusions/8 weeks compared to pretreatment transfusion number in previous 8 weeks. Only RBC transfusions given for Hgb of ≤9.0 g/dL pretreatment will count in RBC transfusion response evaluation. 2)Platelet response (pretreatment,<100x10^9/L):Absolute increase of ≥30x10^9/L for participants starting->20x10^9/L platelets, increase <20x10^9/L to >20x10^9/L by at least 100%. 3)Neutrophil response (pretreatment,<1.0x10^9/L):At least 100% increase and an absolute increase >0.5x10^9/L. 4)Progression or relapse after HI:At least 1 of following: 50% decrement from maximum response levels in granulocytes or platelets, or reduction in Hgb by ≥1.5 g/dL, or transfusion dependence.
Time Frame: as for outcome 1
Population: Safety population was defined as all participants who received any amount of alisertib.
Measure: Number; unit: percentage of participants
Arm/Group | Alisertib 50 mg (Myelodysplastic Syndrome)
Number analyzed (Participants) | 11
percentage of participants
  Erythroid Response | 0
  Platelet Response | 0
  Neutrophil Response | 0
  Progression or Relapse | 0
  Not Available | 91
  Unable to Assess | 9

5. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Deaths
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event. Relationship of each AE to study drug was determined by the Investigator.
Time Frame: First dose of study drug to 30 days after last dose (Up to 18.9 months)
Population: Safety population was defined as all participants who received any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Alisertib 50 mg (Acute Myeloid Leukemia) | Alisertib 50 mg (Myelodysplastic Syndrome)
Number analyzed (Participants) | 46 | 11
participants
  AE | 46 | 11
  SAE | 36 | 8
  Deaths | 20 | 2

6. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as Treatment-Emergent Adverse Events
Description: Vital signs measurements (blood pressure, heart rate, and oral temperature) were obtained throughout the study. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: First dose of study drug to 30 days after last dose (Up to 18.9 months)
Population: Safety population was defined as all participants who received any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Alisertib 50 mg (Acute Myeloid Leukemia) | Alisertib 50 mg (Myelodysplastic Syndrome)
Number analyzed (Participants) | 46 | 11
participants
  Dyspnoea | 12 | 2
  Pyrexia | 10 | 2
  Hypotension | 8 | 0
  Atrial fibrillation | 4 | 1
  Tachycardia | 3 | 0
  Dyspnoea exertional | 2 | 1
  Hypertension | 1 | 1
  Supraventricular tachycardia | 2 | 0
  Weight decreased | 2 | 0
  Tachypnoea | 1 | 0
  Hyperthermia | 1 | 0
  Hypothermia | 1 | 0
  Bradycardia | 0 | 1
  Ventricular tachycardia | 1 | 0

7. Secondary Outcome: Number of Participants With Abnormal Laboratory Values Reported as Treatment-Emergent Adverse Events
Description: Abnormal Laboratory Values for Chemistry or Hematology tests that were assessed by the investigator to be Grade 3 or higher using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE). Grade 3=severe, Grade 4=life threatening or disabling and Grade 5=Death. A treatment--emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: First dose of study drug to 30 days after last dose (Up to 18.9 months)
Population: Safety population was defined as all participants who received any amount of alisertib.
Measure: Number; unit: participants
Arm/Group | Alisertib 50 mg (Acute Myeloid Leukemia) | Alisertib 50 mg (Myelodysplastic Syndrome)
Number analyzed (Participants) | 46 | 11
participants
  Febrile neutropenia | 17 | 4
  Anaemia | 14 | 3
  Thrombocytopenia | 9 | 2
  Neutropenia | 5 | 3
  Leukopenia | 3 | 2
  Hypoalbuminaemia | 4 | 0
  Leukocytosis | 3 | 0
  Hypokalaemia | 3 | 0
  Hyponatraemia | 3 | 0
  Neutrophil count decreased | 3 | 0
  Hypocalcaemia | 2 | 0
  Clostridium difficile colitis | 2 | 0
  Febrile bone marrow aplasia | 1 | 0
  Hypoxia | 1 | 0
  Hyperkalaemia | 1 | 0
  Hypernatraemia | 1 | 0
  Hyperglycaemia | 1 | 0
  Hypoglycaemia | 1 | 0
  Hypomagnesaemia | 0 | 1
  Hypophospataemia | 1 | 0
  Alanine aminotransferase increased | 0 | 1
  Blood bilirubin increased | 1 | 0
  Oxygen saturation decreased | 1 | 0
  Blood culture positive | 1 | 0
  Blood magnesium decreased | 1 | 0
  Blood creatinine increased | 1 | 0
  White blood cell count decreased | 1 | 0
  Gilbert's syndrome | 1 | 0
  Lymphoedema | 1 | 0
  Platelet count decreased | 1 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days after last dose (Up to 18.9 Months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alisertib 50 mg (Acute Myeloid Leukemia) | Alisertib 50 mg (Myelodysplastic Syndrome)
Serious Adverse Events (participants affected / at risk) | 36/46 | 8/11
Other Adverse Events (participants affected / at risk) | 45/46 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib 50 mg (Acute Myeloid Leukemia) (N=46) | Alisertib 50 mg (Myelodysplastic Syndrome) (N=11)
Febrile neutropenia (Blood and lymphatic system disorders) | 13 | 4
Sepsis (Infections and infestations) | 5 | 2
Disease progression (General disorders) | 4 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Pneumonia (Infections and infestations) | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Fatigue (General disorders) | 1 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Serratia bacteraemia (Infections and infestations) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib 50 mg (Acute Myeloid Leukemia) (N=46) | Alisertib 50 mg (Myelodysplastic Syndrome) (N=11)
Fatigue (General disorders) | 15 | 5
Oedema peripheral (General disorders) | 12 | 0
Pyrexia (General disorders) | 9 | 2
Asthenia (General disorders) | 8 | 1
Chills (General disorders) | 6 | 1
Axillary pain (General disorders) | 0 | 1
Catheter site erythema (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 21 | 2
Nausea (Gastrointestinal disorders) | 19 | 3
Stomatitis (Gastrointestinal disorders) | 13 | 4
Vomiting (Gastrointestinal disorders) | 8 | 2
Dysphagia (Gastrointestinal disorders) | 6 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Gingival bleeding (Gastrointestinal disorders) | 4 | 0
Oral pain (Gastrointestinal disorders) | 4 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 1
Proctalgia (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Tongue ulceration (Gastrointestinal disorders) | 1 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 4
Petechiae (Skin and subcutaneous tissue disorders) | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 10 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 2
Neutropenia (Blood and lymphatic system disorders) | 5 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 2
Leukocytosis (Blood and lymphatic system disorders) | 3 | 0
Somnolence (Nervous system disorders) | 11 | 2
Headache (Nervous system disorders) | 5 | 2
Balance disorder (Nervous system disorders) | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Subdural hygroma (Nervous system disorders) | 0 | 1
Oral herpes (Infections and infestations) | 4 | 1
Cellulitis (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 0 | 1
Aspergillosis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 8 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 7 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 0
Tachycardia (Cardiac disorders) | 3 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 4 | 0
Confusional state (Psychiatric disorders) | 2 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 3
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 3 | 0
Haematuria (Renal and urinary disorders) | 3 | 0
Vision blurred (Eye disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Abdominal pain (Gastrointestinal disorders) | 11 | 2
Dizziness (Nervous system disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.